CLINICAL TRIAL: NCT05919017
Title: Exploring the Pharmacokinetic Characteristics of Different Doses of Naltrexone Implants in Patients With Alcohol Use Disorders
Brief Title: Exploring the PK of Different Doses of Naltrexone in Patients With AUD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Sciencare Medical Industries Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ShenzhenSciencare
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: AUD
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo implant, subcutaneous abdominal implant, single dose, 10 placebo tablets implanted
  Interventions: Drug: Placebo
- Naltrexone implant 0.9 g (Experimental): Naltrexone implant, abdominal subcutaneous implantation, single administration, implantation dose is 0.9g (6 naltrexone implants+4 placebo tablets)
  Interventions: Drug: Naltrexone implant
- Naltrexone implant 1.5 g (Experimental): Naltrexone implant, abdominal subcutaneous implantation, single dose of 1.5g (10 naltrexone implants)
  Interventions: Drug: Naltrexone implant

INTERVENTIONS:
Drug: Naltrexone implant — Naltrexone implant
  Arms: Naltrexone implant 0.9 g; Naltrexone implant 1.5 g
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Study Design This study is related to a multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of different doses of naltrexone implants in the treatment of patients with alcohol use disorders (protocol No.: SK2007-NQT-201, hereinafter referred to as II). This study plans to include 60 patients who are interested in participating in this study in Phase II patients, collect PK blood samples from patients, and conduct PK characteristic analysis. The collected plasma samples will be temporarily stored in a -80 ℃ refrigerator and tested after unblinding in Phase II.

DETAILED DESCRIPTION:
Research Design

This study is related to "a multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of different doses of naltrexone implants in the treatment of patients with alcohol use disorders" (protocol No.: SK2007-NQT-201, hereinafter referred to as II). This study plans to include 60 patients who are interested in participating in this study in Phase II patients, collect PK blood samples from patients, and conduct PK characteristic analysis. The collected plasma samples will be temporarily stored in a -80 ℃ refrigerator and tested after unblinding in Phase II.

Research process and PK blood collection

Twelve blood samples were collected from each patient, about 4mL of venous blood were collected 0 h before administration (within 4h before administration) and 4h, 12h, D1 (24h), D7, D14, D28, D56, D84, D112, D140, D168 days after administration.

At the planned blood collection point, collect approximately 4mL of blood sample into a labeled heparin sodium anticoagulant vacuum collection vessel. After collecting each tube of blood, gently invert it back and forth immediately and pay attention to hemolysis to fully mix the blood with anticoagulants to ensure anticoagulant effect. After sample collection and before centrifugation, the blood sample needs to be placed upright in an ice water bath and transported to the sample pretreatment room. Within 1 hour, the blood sample should be placed in a low-temperature centrifuge for centrifugation.

ELIGIBILITY:
Selection criteria:

1. Volunteer to participate in clinical research; Fully understand and be informed of this experiment and sign informed consent; Willing to follow and capable of completing all testing procedures;
2. The age at the time of signing the informed consent form is ≥ 18 years old;
3. Patients diagnosed as moderate to severe alcohol use disorders based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) (four or more items that meet the diagnostic criteria);
4. Have completed withdrawal treatment and have no obvious alcohol withdrawal symptoms for at least one week (≥ 7 days) before randomization/administration [Clinical Institute Alcohol Dependence Withdrawal Assessment Form (CIWA-Ar) score<7 points];
5. Able to provide TLFB alcohol consumption information 2 weeks prior to withdrawal and/or screening;
6. During the 4-week period before withdrawal and/or screening, drink heavily at least twice a week;

Qualified subjects of childbearing age (male and female) must agree to take effective contraceptive measures (hormone or barrier therapy or abstinence) with their partners during the trial period.

Exclusion criteria:

Participants who meet any of the following criteria cannot be selected for the experiment:

1. The researcher determines that participating in this experiment does not comply with the rights and interests of the subjects, or any other circumstances that do not allow the subjects to conduct the study safely;
2. Pregnant and reproductive age women with positive pregnancy tests or lactating women, including those who planned to conceive during the study period. Note: Here, women of childbearing age refer to women with fertility. The following criteria must be met, regardless of their sexual orientation or whether they have undergone tubal ligation: 1) have not undergone hysterectomy or bilateral ovariectomy; Or 2) Have not experienced natural menopause for more than 12 consecutive months (i.e., have menstruated at any time during the previous 12 consecutive months);
3. Significant abnormalities in liver function (such as AST or ALT exceeding twice the upper limit of normal values) or liver failure (including but not limited to: abdominal fluid accumulation, prolonged prothrombin time, international standard ratio (INR) ≥ 1.7, esophageal varicose disease) or liver and gallbladder ultrasound display results have a significant impact on the judgment of the efficacy and safety of the study drug;
4. Suffering from uncontrollable active infectious diseases in clinical practice, such as active hepatitis B (positive for hepatitis B surface antigen (HBsAg) detection and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) copy number>1000 IU/ml), active hepatitis C (positive for hepatitis C virus antibody and hepatitis C virus (HCV) ribonucleic acid (RNA)), etc;
5. A history of congenital hemorrhagic disease (such as hemophilia) or any clinically significant bleeding, or abnormal platelet function, or prothrombin time (PT) exceeding the upper limit of normal values by more than 3 seconds (sec) during coagulation function testing, or platelet count<50 × 109/L；
6. Previous history of severe pancreatitis or severe tremor delirium episodes;
7. According to the judgment of the researchers, the subjects have any severe/uncontrollable systemic diseases (such as respiratory, circulatory, digestive, nervous, hematological, urogenital, endocrine system diseases) or mental illnesses (such as severe depression, schizophrenia, bipolar disorder, etc.) or other major diseases that the researchers believe will hinder the provision of informed consent and make participation in the study unsafe Complicating the interpretation of research outcome data or otherwise affecting the achievement of research objectives;
8. Hospitalization or surgery may be required during the study period, including planned elective surgery or hospitalization that cannot be postponed;
9. According to the DSM-5 standard, currently diagnosed (within one year prior to randomization/administration) with substance use disorders other than alcohol, such as benzodiazepines, amphetamines, opioids, or cocaine;
10. Within 30 days before randomization/administration, I have taken drugs to prevent relapse (such as naltrexone) or received systematic psychological support treatment;
11. Currently undergoing treatment for opioid, amphetamine, alcohol, and other substance use disorders, or receiving opioid treatment within 7 days before randomization/administration, opioid treatment may be required during the study period, or on the day of randomization/administration, urine opioid, marijuana, amphetamine, and other drugs tested positive or naloxone challenge test positive;
12. Allergies to research drugs or their excipients (polylactic acid, magnesium stearate), local anesthetics;
13. Participating in any study drug or device research, or having used any study drug or device within 30 days prior to randomization/administration;
14. If there is a skin infection or systemic skin disease at the site of implantation surgery, it is determined that it can affect the effectiveness and safety evaluation of the study drug;
15. Clinical or laboratory evidence suggests that human immunodeficiency virus (HIV) or syphilis are carried/infected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | 168 day
  PK
AUC | 168 day
  PK

CONTACTS AND LOCATIONS:
Overall Officials: zou xuhui, Dr, Principal Investigator — Hunan Second People's Hospital
Locations (1):
- Hunan Second People's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No